CLINICAL TRIAL: NCT04692922
Title: Prognostication of Recovery in Early Disorders of Consciousness Study
Acronym: PREDICT
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2020P002706
Record Dates: First submitted 2020-11-10; First posted 2021-01-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Disorders of Consciousness Due to Severe Brain Injury
Keywords: Disorders of consciousness; Advanced neuroimaging; Neuroprognostication
MeSH Terms: conditions — Consciousness Disorders | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with disorders of consciousness: patients with a diagnosis of coma, vegetative state, or minimally conscious state minus (i.e. minimally conscious state without language function)
  Interventions: Diagnostic Test: MRI; Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: MRI — MRI will include structural sequences (e.g., T1 weighted imaging, T2 weighted imaging, T2 FLAIR, diffusion weighted imaging with apparent diffusion coefficient, susceptibility weighted imaging, and diffusion tensor imaging). Using the structural sequences we will make note of the types of brain lesions (e.g., ischemic stroke, hemorrhage, hypoxic-ischemic brain injury), and the locations of these brain lesions. MRI will also include fMRI under three conditions: while the patient is at rest (to evaluate resting state functional connectivity), while the patient is exposed to auditory stimuli (to evaluate passive fMRI responses to stimuli), and while the patient is asked to follow commands (to evaluate active fMRI responses to tasks).
Diagnostic Test: EEG — The EEG will include resting, stimulus-based, and task-based assessments of brain function.

SUMMARY:
By collecting multimodal metrics (e.g., clinical factors, neuroimaging, and EEG) in the early phase of severe brain injury (i.e., during the acute hospitalization when a patient has impaired consciousness), and measuring the patients' recovery of consciousness, function, and quality of life in the late phase (at 6 months following the brain injury), we aim to construct an algorithm that synthesizes the results of these metrics to help predict recovery.

DETAILED DESCRIPTION:
The primary aim of this research proposal is as follows: By collecting multimodal metrics (e.g., clinical factors, neuroimaging, and EEG) in the early phase of severe brain injury (i.e., during the acute hospitalization when a patient has impaired consciousness), and measuring the patients' recovery of consciousness, function, and quality of life in the late phase (at 3, 6, and 12 months following the brain injury), we aim to construct an algorithm that synthesizes the results of these metrics to help predict recovery.

There will also be secondary aims as follows:

1. To identify patient phenotypes with predictive significance, in order to revise our classification scheme for disorders of consciousness in a clinically meaningful and data driven manner.
2. To compare prognostic value between metrics.
3. To determine how the initial goals of care expressed in the acute setting (i.e., the expected quality of life associated with disability) compare to the actual quality of life in the chronic setting (i.e., the actual quality of life associated with disability).
4. To compare the prognostic value of metrics between different etiologies of brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Acute brain injury (including ischemic stroke, intracranial hemorrhage, anoxic brain injury, traumatic brain injury, encephalitis)
* Inability to follow commands, speak intelligibly, or communicate (i.e., diagnosis of coma, vegetative state, or minimally conscious state minus) due to the underlying brain injury and within 28 days of the brain injury
* Age 18 or greater.

Exclusion Criteria:

* Subjects will be excluded if they do not speak English (given the reliance on verbal questionnaires conducted in English) or if they regain the ability to follow commands, speak intelligibly or communicate (i.e., improves to minimally conscious state plus or greater) before they undergo MRI or EEG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disorders of consciousness following acute brain injury
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended | 6 months following enrollment
  Metric of neurologic function. The minimum score is 1, and the maximum score is 8. Higher scores represent less disability (8 represents non-disabling symptoms, 1 represents death).

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Edlow, MD, Principal Investigator — Massachusetts General Hospital